CLINICAL TRIAL: NCT04369989
Title: Observational Study of COVID-19 Treatment Efficacy
Status: Terminated | Type: Observational
Why Stopped: Review of data revealed poor correlation with hypothesis and data quality challenges.
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, David Hall, Senior Vice President Information Systems / Chief Information Officer, Integrated Solutions, OSF Healthcare System
Other Study IDs: 1589936
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Coronavirus; Coronavirus Infection; Corona Virus Infection; COVID; Sars-CoV2; Coronavirus as the Cause of Diseases Classified Elsewhere; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere; COVID-19; Coronavirus Disease; Coronavirus Sars-Associated as Cause of Disease Classified Elsewhere
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hydroxychloroquine - NO: Did not receive / are not receiving any Hydroxychloroquine
  Interventions: Other: No intervention
- Hydroxychloroquine - YES - started before: Hydroxychloroquine date started was before the date recorded for signs of respiratory distress
  Interventions: Other: No intervention
- Hydroxychloroquine - YES - started same: Hydroxychloroquine date started was the same as the date recorded for signs of respiratory distress
  Interventions: Other: No intervention
- Hydroxychloroquine - YES - started after: Hydroxychloroquine date started was after the date recorded for signs of respiratory distress
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To compare various treatments provided to positive COVID-19 patients at locations across the OSF Ministry. Provide the opportunity to compare the effectiveness of various treatments and treatment timelines provided to specific cohorts of patients that have the potential to impact future treatment plans for COVID-19 patients and/or future research hypotheses.

DETAILED DESCRIPTION:
Background:

Several studies have indicated a potential role for Hydroxychloroquine in the treatment of COVID-19 as caused by the SARS-CoV-2 virus. Hydroxychloroquine has demonstrated potent inhibition of SARS-CoV-2 in vitro. Hydroxychloroquine and azithromycin together have significantly reduced SARS-CoV-2 viral carriage over 6 days compared to a placebo and COVID-19 patients who received a 5 day regimen of 400mg/day of Hydroxychloroquine had significantly shortened times to clinical recovery characterized by improved pneumonia compared with patients who did not receive Hydroxychloroquine.

Within OSF Healthcare approximately 50% of SARS-CoV-2 infected patients are currently receiving some form of Hydroxychloroquine during the course of their hospitalization. The utilization of this treatment has been approved by the FDA based upon the limited data available.

Significance:

The optimal treatment regimen for COVID-19 patients has yet to be defined. Several small studies have indicated a potential role for the utilization of Hydroxychloroquine in the treatment of SARS-CoV-2 infected patients. However, very little evidence exists around the optimal treatment regimen and efficacy with regard to tangible outcomes. This observational retrospective/prospective chart review study aims to help provide epidemiological data that may help to provide guidance to clinicians for both future patients, as well as provide clinicians guidance for study design of more definitive controlled studies. Given the rapid spread of this disease, the high mortality rate associated with it and the impact of the disease upon society this study is anticipated to have the potential to contribute significantly to the treatment of SARS-CoV-2 infected patients.

Study Design and Methodology:

The study will be a retrospective/prospective observational study of cohorts of hospitalized patients across the OSF Healthcare System who have tested positive for SARS-CoV-2 and exhibit signs or symptoms of respiratory distress during the course of their hospitalization. The outcomes of patients who both receive and do not receive Hydroxychloroquine will be compared, with particular attention to the timing of administration in relationship to the onset of respiratory distress. Respiratory distress will be defined as a low SpO2, an elevated respiratory rate or an increased oxygen demand. Hydroxychloroquine administration will be defined as a documented administration of the medication on the patient's medication administration record (MAR). Administration of Hydroxychloroquine prior to the onset of respiratory distress, administration of Hydroxychloroquine on the day of respiratory distress and administration of Hydroxychloroquine following the onset of respiratory distress will all be assessed and compared across three outcome metrics; progression to an ICU location of care, progression to ventilator support and mortality.

* Patients at all OSF HealthCare locations across the Ministry that meet Inclusion/Exclusion criteria will be cohorted by:

  * Hydroxychloroquine administered - yes (including the date started)
  * Hydroxychloroquine - no
* For the Hydroxychloroquine administered - yes cohort, further subdivide into 3 cohorts:

  * Hydroxychloroquine date started was before the date recorded for signs of respiratory distress
  * Hydroxychloroquine date started was the same as the date recorded for signs of respiratory distress
  * Hydroxychloroquine date started was after the date recorded for signs of respiratory distress
* At this point the investigators would have 4 cohorts:

  * Hydroxychloroquine - No
  * Hydroxychloroquine date started was before the date recorded for signs of respiratory distress
  * Hydroxychloroquine date started was the same as the date recorded for signs of respiratory distress
  * Hydroxychloroquine date started was after the date recorded for signs of respiratory distress
* These 4 cohorts would be compared to determine any difference in the following metrics:

  * Mortality
  * ICU Admissions
  * Ventilator use
* Additional study of additional treatment regimens using a similar design may be repeated for the following treatments

  * Hydroxychloroquine + Azithromycin
  * Remdesivir (This is a compassionate use medication with very limited use in OSF. Observational study of this would be significantly limited and therefore unlikely to be undertaken)
  * Non-steroidal anti-inflammatories (some indication that these lead to poorer outcomes)

Study Procedures:

OSF Data Analytics will pull reports of confirmed positive COVID-19 subjects. The data will be kept securely on password-protected computers and analyzed by applicable research personnel listed on this study.

Data Use and Management:

1. Results of this study will be presented within OSF Healthcare at national meetings and/or published in academic journals. The investigators will not disclose any subject PHI or identifying personal information in any presentation or publication about the study.
2. The study investigators will be responsible for data safety monitoring. This is an observational study which only involves data collection from the hospital/institutional sources (e.g., hospital notes, office visit notes,). This study does not dictate any specific surgical treatments or medications. All procedures performed on the patients are standard of care and the study does not involve any additional hospital visits for subject or the parents/guardians. Data that will be collected from patient records will be securely stored on password-protected computers accessible only by applicable research personnel.

Data Analysis:

Data analysis will be performed by the PI and applicable research personnel.

Oversight and Ethics:

This study will be conducted in compliance with the Peoria IRB research policies and procedures and all applicable laws and regulations. The staff members will perform the study in accordance with the protocol, and will report unexpected problems in accordance with the Peoria IRB policies and procedures and applicable laws and regulations. Collection, recording, and reporting of data will be accurate and will ensure the privacy, health, and welfare of research subjects during and after the study.

Privacy and Confidentiality:

Study staff will maintain the highest degree of confidentiality permitted for clinical and research information obtained from the participants. Medical and records will be maintained in the strictest confidence. However, as a part of the quality assurance and legal responsibilities of an investigation, the clinical site must permit monitoring representatives of various governing facilities to examine clinical records for the purpose of quality assurance reviews, audits, and evaluations of the registry safety and progress. Unless required by the laws that permit copying of records, only the coded identity associated with documents or with other participant data may be copied (and all personally identifying information must be obscured). Authorized representatives as noted above are bound to maintain the strict confidentiality of medical and research information that is linked to individuals. The clinical site will normally be notified before auditing visits occur.

Risks:

The main risk in this study is the potential breach of privacy and loss of confidentiality. There is minimal risk of likelihood of harm. All reasonable safeguards to secure the confidentiality of information will be taken by the investigators and their research personnel.

ELIGIBILITY:
Inclusion Criteria:

* test positive for COVID-19
* be inpatient
* Have signs of respiratory distress = had either an SpO2 of less 95% or lower recorded or a respiratory rate RR >20 (21 or more) recorded and <60 (eliminate aberrant charting)

Exclusion Criteria:

* Age less than 18
* Currently actively in an investigational drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at all OSF HealthCare locations across the OSF Ministry that meet inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Mortality during the COVID-19 treatment hospital encounter | up to 6 weeks
ICU admission during the COVID-19 treatment hospital encounter | up to 6 weeks
Ventilator use during the COVID-19 treatment hospital encounter | up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- OSF HealthCare St Francis Medical Center, Peoria, Illinois, United States

REFERENCES:
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Efficacy of hydroxychloroquine in patients with COVID-19: results of a randomized clinical trial Zhaowei Chen, Jijia Hu, Zongwei Zhang, Shan Jiang, Shoumeng Han, Dandan Yan, Ruhong Zhuang, Ben Hu and Zhan Zhang; medRxiv preprint doi: https://doi.org/10.1101/2020.03.22.20040758. 03.31.2020